CLINICAL TRIAL: NCT00346866
Title: Anecortave Acetate Versus Placebo in AMD Patients Following PDT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-00-07
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: AMD
MeSH Terms: interventions — anecortave acetate

INTERVENTIONS:
Drug: anecortave acetate

SUMMARY:
The purpose of this study was to evaluate the efficacy of anecortave acetate for depot suspension (30 mg and 15 mg) plus PDT versus PDT alone with respect to maintenance of visual acuity in patients with wet AMD.

ELIGIBILITY:
Inclusion Criteria:

* AMD disease

Exclusion Criteria:

* Age

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136
Dates: Start 2000-05; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Mean change from the baseline in logMAR visual acuity score at Month 6

SECONDARY OUTCOMES:
% patients who maintained vision, number of months of angiographic evidence of needing PDT re-treatment, and mean lesion sizes for the total choroidal neovascularization (CNV) and the classic component to the total CNV.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Zilliox, Study Director — Alcon Research
Locations (1):
- Facility, Beachwood, Ohio, United States